CLINICAL TRIAL: NCT02444403
Title: Proyecto ESCUDO: Police Training to Reduce Occupational Needlesticks and HIV Among Substance Users
Brief Title: Police Training to Reduce Occupational Needlesticks and HIV Among Substance Users
Acronym: ESCUDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Open Society Foundations (Unknown); UCSD Center for AIDS Research (CFAR) (Unknown); Mexico-U.S. Border Health Commission, Mexico section (Unknown)
Responsible Party: Principal Investigator, Steffanie Strathdee, Associate Dean of Global Health Sciences, Harold Simon Professor, Chief, Division of Global Public Health, University of California San Diego, Department of Medicine, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01DA039073 (NIH)
Record Dates: First submitted 2015-05-12; First posted 2015-05-14 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Occupational Needlestick Injuries
Keywords: HIV; Viral hepatitis; HCV; Needle-stick injury; Needle/syringes; Structural intervention; Stepped wedge; Police; Occupational safety; Police Training
MeSH Terms: conditions — Needlestick Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Police Education Program (PEP) (Other): The entire police force mandated for periodic refresher training will be assigned to classes which receive one PEP course over 2 years.
  Interventions: Behavioral: Police Education Program designed to align law enforcement and HIV prevention in Tijuana

INTERVENTIONS:
Behavioral: Police Education Program designed to align law enforcement and HIV prevention in Tijuana — The 3.5-hour PEP course consists of 3 modules. Module I covers basic epidemiology, prevention and treatment of HIV, viral hepatitis and STIs, safe syringe disposal and fundamentals of addiction. Post-exposure protocols and appropriate follow-up procedures are outlined. Module II covers key provisions of Mexico's national drug policy (narcomenudeo, which defines amounts of drugs allowed for personal possession), as well as other legal provisions pertinent to HIV prevention, including the legality of syringe and condom possession. Module III covers public health-based interventions targeting PWID (SEPs, OST) and deconstructs myths typical among law enforcement (i.e., drug users do not care about their health, SEPs increase the risk of NSIs).
  A sub-cohort sample will be invited to undergo pre- and post-PEP surveys with semi-annual follow-up for 2 years to assess self-reported NSIs (Aim 1), attitudinal and behavior changes (Aim 2) and mediators/moderators (Aim 3).
  Other Names: Police Education Program (PEP)

SUMMARY:
Background: Policing practices are key drivers of HIV among people who inject drugs (PWID). This study prospectively examines the impact of a police education program (PEP) to align law enforcement and HIV prevention. PEPs incorporating HIV prevention, (including harm reduction programs like syringe exchange) have been successfully piloted in several countries but were limited to brief pre-post assessments; the impact of PEPs on policing behaviors and occupational safety is unknown. Objectives: Proyecto ESCUDO (Project SHIELD) aims to evaluate the efficacy of the PEP on uptake of occupational safety procedures, as assessed through the incidence of needle stick injuries (NSIs) (primary outcome) and changes in knowledge of transmission, prevention and treatment of HIV and viral hepatitis; attitudes towards PWID, adverse behaviors that interfere with HIV prevention, and protective behaviors (secondary outcomes). The investigators hypothesize that, over the course of the 24-month follow-up, the PEP will be associated with significant declines in NSI incidence, improved knowledge of HIV and related infections, uptake of occupational safety measures, and decreases in behaviors that undermine HIV prevention (e.g. syringe confiscation, police harassment of PWID at opioid substitution therapy and syringe exchange programs). Methods/Design: ESCUDO is a Hybrid Type 2 design that simultaneously tests an intervention and an implementation strategy. Using a modified stepped-wedge design involving all active duty street-level police officers in Tijuana (N= ~1200), the investigators will administer one 3-hour PEP course to groups of 20-50 officers until the entire force is trained. NSI incidence and geo-coded arrest data will be assessed from department-wide de-identified data. Of consenting police officers, a sub-cohort (N=500) will be randomly sampled from each class to undergo pre- and post-PEP surveys with semi-annual follow-up for 2 years to assess self-reported NSIs, attitudes and behavior changes. Impact on PWIDs will be externally validated through a parallel cohort of Tijuana PWIDs. Discussion: This is the first trial to assess efficacy of a PEP on policing behaviors that place PWID and police at elevated risk of HIV and blood-borne infections. Findings may help bring PEPs to scale in the growing number of countries where policing is a documented driver of HIV acquisition.

DETAILED DESCRIPTION:
The Police Education Program (PEP) and its evaluation component, has been titled Proyecto ESCUDO (Project SHIELD). This project has the following aims: 1) To evaluate the efficacy of the PEP on uptake of occupational safety procedures, as assessed through the incidence of occupational needle-stick injury (NSI) (primary outcome), monitored by a department-wide NSI surveillance program, and self-reported NSI; 2) To evaluate the efficacy of the PEP on changes in the following secondary outcomes: i) knowledge of transmission, prevention and treatment of HIV and related infections (sexually transmitted infections (STIs) and viral hepatitis); ii) attitudes towards people who inject drugs (PWID); iii) adverse behaviors that interfere with HIV prevention (i.e., arrests near syringe exchange programs (SEP) and drug treatment locations); iv) protective behaviors (e.g., use of barrier protection, self-reported reductions in syringe confiscation). 3) To assess potential mediating and moderating factors that influence PEP efficacy, including changes in knowledge and attitudinal factors and occupational constructs. The investigators hypothesize that, over the course of the 24-month follow-up, the PEP will be associated with significant declines in NSI incidence, improved knowledge of HIV and related infections, uptake of occupational safety measures, and decreases in behaviors that undermine HIV prevention (e.g. syringe confiscation, police harassment of PWID at opioid substitution therapy (OST) and SEPs).

Hypotheses:

H1. The PEP will be associated with a significant decline in NSI incidence among the force during follow-up.

H2.1. The PEP will be associated with significantly increased knowledge of transmission, prevention and treatment of HIV and HCV among Tijuana police officers participating in the sub-cohort.

H2.2. The PEP will be associated with significant improvements in attitudes towards PWID, sex workers and HIV-infected persons.

H2.3. The PEP will be associated with significantly fewer reports of syringe confiscation by police officers.

H2.4. The PEP will be associated with lower incidence of arrests near SEP and drug treatment locations.

H2.5 The PEP will be associated with increased use of barrier protection during pat-downs and arrests.

H2.6. The PEP will be associated with increased knowledge about the narcomenudeo drug policy reform.

H3.1 The impact of PEP on NSI incidence and adverse and protective behaviors will be moderated by officers' motivation to undergo the training, years in the force, and autonomous support received from supervisors.

Conceptual Framework of the PEP: The trans-contextual Model (TCM) has been successfully used to evaluate injury prevention PEPs in international settings (Chung-Chan and Hagger 2012). The investigators applied the TCM to conceptualize and assess mechanisms through which the PEP can impact occupational safety and officers' behaviors. This model incorporates key theoretical constructs from self-determination theory (SDT) (Deci and Ryan 2000) and the theory of planned behavior (TPB) (Ajzen 1991). TPB emphasizes the role of psychosocial factors in affecting decision making processes that translate to changes in behavior. Herein, such factors include trainee attitudes, subjective norms, self-efficacy, and intentions. These TPB constructs have had robust predictive value in the realm of injury prevention (Sheeran and Silverman 2003, Lajunen and Rasanen 2004). SDT highlights the role of motivation and perceived autonomy as "regulators" that may mediate the impact of training initiatives on trainee practices and adherence. Perceived support by supervisors (autonomy support) for injury prevention (Chan, Lonsdale et al. 1977) and motivation to participate in an educational intervention are known antecedents for change in behavioral and corollary endpoints (Standage, Duda et al. 2005). Validated in the realm of occupational safety and injury prevention (Chan and Hagger 2012, Hagger and Chatzisarantis 2012), TCM is based on the complex interplay between SDT and TPB factors in shaping the impact of educational interventions (Chung-Chan and Hagger 2012). The TCM model also suggests that changes in self-efficacy produced by training can be transferred to domains that are related, but do not serve as the focus of the training intervention (Chung-Chan and Hagger 2012). Herein, TCM elucidates the pathways through which the PEP may shift ancillary police activities, including adherence to departmental procedures and drug policies (e.g. targeting PWID for enforcement activities as they seek to access SEPs or OST). These shifts may improve police occupational safety by reducing the prevalence of adverse encounters with PWID, but they may also have collateral population health benefits such as reducing risk behavior and infectious disease incidence among PWID. TCM has been widely used in the context of physical education training (Hagger, Chatzisarantis et al. 2003, Hagger, Chatzisarantis et al. 2005, Pihu, Hein et al. 2008, Hagger, Chatzisarantis et al. 2009), and research on police occupational health, but its use in the assessment of a PEP focused on NSI prevention is innovative (Chung-Chan and Hagger 2012).

PEP Intervention: Based on best practices established by Beletsky et al (Davis and Beletsky 2009, Beletsky, Agrawal et al. 2011, Silverman, Davis et al. 2012, Beletsky, Thomas et al. 2013), and with active input from the Instituto de Capacitacion y Adiestramiento Profesional (ICAP, Tijuana Police Academy) instructional experts, the investigators culturally and linguistically adapted existing PEP materials that bundle occupational safety information with content addressing the legal, scientific, and logistical underpinnings of HIV prevention. Through train-the-trainer workshops, the investigators prepared ICAP instructors by building knowledge, pedagogical skills and capacity, with an emphasis on a peer-to-peer perspective to maximize uptake (Davis and Beletsky 2009). An initial team of three trained ICAP instructors will deliver the standardized curriculum through slide-assisted oral presentations in one-hour sections (i.e. modules), offered consecutively in a single session. The entire training lasts approximately three-and-a-half hours. The entire police force mandated for periodic refresher training will be assigned to classes which receive one PEP course over 2 years.

Study Design: ESCUDO is a Hybrid Type 2 design that simultaneously tests an intervention and an implementation strategy (Curran, Bauer et al. 2012 ). This study has three levels: 1) Implementation of the PEP across the entire Tijuana police department using a stepped wedge design, and evaluating department-wide NSI incidence for the primary study outcome; 2) Prospective 24-month follow-up of a random sub-cohort of police officers sampled from each PEP class to assess behavioral outcomes; 3) Simultaneous longitudinal follow-up of a parallel cohort of PWID to independently assess their experiences with police. Each of these components is described below.

Level 1: Implementation of the PEP across the Tijuana Police Department. ESCUDO was initially conceived as a modified stepped-wedge randomized controlled trial involving staggered roll-out of the PEP where participants are randomly selected to transition from the control to intervention in classes of equal numbers over a two year period. However, since randomly assigning officers to PEP classes would interfere with the department's programmatic priorities, the investigators modified the design to integrate the PEP into regularly scheduled refresher training classes that were being held for other purposes (e.g., basic police tactics). The design the investigators adopted maintains core features of a stepped wedge design, whereby the pre-intervention period for each officer is treated as the control. On a weekly basis, one cluster (i.e., class of 20-50 officers from different ranks and precincts undergoing regularly scheduled refresher training) will 'step up' and cross over from the control to the intervention condition by receiving PEP training, until the entire force of 1200 street-level officers is trained. Incidence of NSIs (primary outcome, Aim 1) and incidence of arrests near SEPs and drug treatment programs (secondary outcome, Aim 2), will be assessed on the entire police department based on de-identified data.

The primary endpoint of Proyecto ESCUDO is NSI incidence (Aim 1). Since NSIs tend to be under-reported, the investigators will collect these data two ways: 1) Through the NSI Surveillance and Response Program (NSRP) based on prospective data from the entire police department (Level 1); 2) Through the ESCUDO sub-cohort (N=500; Level 2; see below). The first approach utilizes the NSRP that was implemented in 2014 by our team in collaboration with the Police Department and the Office of Municipal Health (DMS) in Tijuana. The NSRP encourages officers experiencing a NSI to notify their direct supervisor and immediately go to the main office of the DMS Department of Legal Medical Experts. These are staffed 24-hours a day by a certified medical doctor in a private medical exam room where they complete an NSI Exposure Report Form detailing the circumstances of exposure. To facilitate reporting of NSIs, the Tijuana police cars have a sticker outlining the NSI protocol, and the State Ministry of Health Office in Tijuana has made free HIV, Hepatitis C, syphilis and Hepatitis B tests available on site. NSI forms will be kept in a locked cabinet on site; the Head of Planning and Special Projects at Tijuana's Police Department will provide quarterly reports to our team and the Data Safety and Monitoring Board including date of NSI, whether the officer had undergone the PEP, date of training, and context of the NSI. No identifiers are included.

Survey Data: Police officers who consent to ESCUDO are given pre and post-PEP surveys that are self-administered. Each survey takes 10-15 minutes to complete. The survey assesses lifetimes and recent on-duty NSIs (Aim 1), and knowledge, attitudes, subjective norms, intentions, self-efficacy for adopting protective behaviors and adverse and protective behaviors affecting NSIs and acquisition of HIV and other blood-borne infections (Aim 2). The survey was adapted from items previously used by Beletsky et al. in domestic and international settings (Davis and Beletsky 2009, Beletsky, Agrawal et al. 2011, Beletsky, Thomas et al. 2013), and piloted in Tijuana. Since knowledge of HIV/AIDS in Tijuana is low (Robertson, Ojeda et al. 2012), the investigators will utilize an 18-item, true/false scale that assesses awareness of HIV symptoms, transmission, and prevention (e.g., "People who have been infected with HIV quickly show serious signs of illness") (Carey and Schroder 2002). The investigators have used this scale in other Tijuana studies (α = 0.75 to 0.89; test-retest reliability= 0.76 to 0.94). Attitudinal, subjective (perceived social) norms, self-efficacy, and intention items developed by Fisher and Fisher will be assessed using a 5-item Likert scales (Strongly agree-strongly disagree) (Fisher, Fisher et al. 1994). Items expressing both positive and negative statements like "Syringe Exchange Programs increase the risk of needle-stick injuries for police" will assess attitudes on vulnerable groups. For subjective norms, statements like "most of my colleagues think it's important to follow official search safety procedures" will be utilized. Self-efficacy for preventive behaviors will be assessed by items like "I am confident that I can prevent on-duty NSIs." To assess intended practices, the investigators will utilize items such as "Next time a suspect informs me that he has a syringe, I will confiscate it." These domains are consistent with central tenets of TPB (Ajzen 1991).

SDT highlights the importance of motivational regulation and autonomy support in evaluating training interventions. To measure motivational constructs, the investigators adopted items from the Perceived Locus of Causality scale and the corollary amotivation subscale (Goudas, Biddle et al. 1994). Items using the stem, 'I am participating in this training because:' will list 4 items per scale. Measures include 'trainings are interesting and fun' (intrinsic motivation; α =.88), 'because occupational safety is important to me' (identified regulation), 'because I am required to do so' (external regulation; α =.81), and 'but I am not interested in this topic' (amotivation; α =.84) (Standage, Duda et al. 2005). Support for these measures is based on diverse training and other intervention evaluation research, including Spanish-speaking settings (Goudas, Biddle et al. 1994, Ntoumanis 2001, Otis and Pelletier 2005, Standage, Duda et al. 2005, Moreno, Cervello et al. 2007). Autonomy support from supervisors will be measured using an adaptation of the Health Care Climate Questionnaire (Baard, Deci et al. 2004), which uses an analogous Likert framework with a series of items such as: ''My supervisor understands me'' (α=.92). Use of these measures is supported by prior research in injury prevention among police (Chung-Chan and Hagger 2012).

Geo-coded Arrest Data: In addition to NSI surveillance data, the Tijuana police department is providing our team with geo-coded arrest data to determine the extent to which the PEP decreases the number of arrests near SEP and OST sites in Tijuana (Aim 2). Based on methodology developed during preliminary studies (Brouwer, Rusch et al. 2012), the investigators will examine spatial overlap between drug-related arrests and SEPs/drug treatment sites using data mapped into GIS-based software, ArcMap 10.1 (ESRI, Redlands, CA). Available drug possession arrest data includes all arrests in which ≥1 charge concerned drug possession over the legal limit, drug-related crimes, the neighborhood (colonia) where the arrest occurred and month of arrest. Using the Getis-Ord Gi* statistic, the investigators will examine spatial patterns to identify hotspots of drug-related arrests at the colonia-level per 1000 adult residents (e.g., neighborhoods with significantly higher or lower rates of arrests than expected if arrests were randomly distributed across space). The investigators will determine whether there was a higher rate of drug-related arrest in colonias with better access to SEPs/OST sites. Access to SEPs/drug treatment sites will be determined by applying a method proposed by Cooper et al (Cooper, des Jarlais et al. 2011) that calculates the percent of a colonia's surface area within a 1350m radius of a SEP/drug treatment site (the 1350m buffer zone corresponds to the median area of colonias in Tijuana). Colonias with no surface area within the buffer zone will be defined as not having access. Further, the investigators examine whether there is a significant increase in the average number of arrests in colonias with greater surface area within the buffer zone through modeling this relationship using Poisson regression.

Level 2: Aim 2 of Proyecto ESCUDO is to determine whether the PEP changes policing behaviors. Therefore, the investigators will assess self-reported NSIs, changes in attitudes about HIV and related infections, attitudes towards PWID, and adverse and protective behaviors that influence blood-borne transmission risks among police and PWID as secondary outcomes among a sub-cohort of police officers sampled from the PEP classes. Specifically, at the beginning of each PEP session, staff will explain to the class of police officers that while the PEP training is mandatory, the ESCUDO evaluation is voluntary. Officers not wishing to participate are told that they can submit blank pre- and post-PEP surveys if they do not wish to disclose their non-participation. A unique identification code will be generated for each officer, based on their day of birth, first initial, first letter of father's last name and mother's last name. Written informed consent to participate in ESCUDO is then obtained for the pre- and post-PEP surveys, as well as a separate consent for follow-up. Only the latter consent asks for personal information to permit study staff to contact them. The consent form for follow-up also asks each officer whether they had ever encountered syringes on duty and in the last 6 months.

Eligibility criteria for the Level 2 component of the study requires that only officers who consent complete the pre- and post-PEP surveys and report encountering syringes within the last 6 months comprise the follow-up sampling frame. To achieve sufficient power the study statistician applies an algorithm to randomly sample approximately 42% of the eligible officers from each class of 20-50 officers who are subsequently contacted for follow-up visits. A total of 500 officers in the sub-cohort will be recruited. This sub-cohort will undergo self-administered surveys pre-PEP, immediately post-PEP and 3, 6-, 12, 18-, and 24-months post-PEP.

While this design has standard features of a stepped wedge design (i.e., staggered transition from the control to intervention), the evaluation differs. Unlike the standard stepped wedge design where every cluster is assessed at each step, only one cluster will be evaluated per step for most secondary outcomes. This was done because it would be impractical to follow 1200 officers for 2 years, and power is sufficient with a sample size of 500 for most outcomes. Unlike the traditional step wedge design where evaluation stops once the last cluster transitions from control to intervention, each member of the sub-cohort will be followed for 2 years.

Follow-Up Survey: While all 1200 police officers are invited to complete the pre-PEP survey and post-PEP survey immediately following the training with informed consent, the post-PEP follow-up interviews occurring at 3, 6, 12, 18 and 24 months post-training are to be conducted exclusively on the sub-cohort (N=500). The above measures will be adapted to focus on the appropriate recall period. Participants will receive a voucher for movie tickets (equivalent 20 USD) for each follow-up interview.

Follow-up: Follow-up interviews will be conducted only among the sub-cohort (N=500), who will be asked to provide locator information at their baseline interview (i.e., home and cell phone, pager, email, address), and ways they prefer to be contacted (e.g., SMS text).

Statistical Analysis (Aims 1-3): The primary analysis will consist of examining outcomes in the pre-PEP vs. post-PEP period utilizing generalized linear mixed models (GLMM) applied to repeated measures analysis of clustered data. Mixed effects models will allow us to adjust for both within-subject and within-cluster correlations; one random effect will capture the within cluster correlation and another will capture the nested subject-within-cluster correlation.

Stepped wedge designs reduce contamination bias, considering that each cluster (here, each class) acts as its own control and hence provides data in both control and intervention periods (Brown and Lilford 2006). Some degree of contamination is likely since PEP classes will occur over 2 years and because of the social nature of policing. The investigators will attempt to measure this by asking officers in the sub-cohort whether other officers had discussed any of the training topics with them prior to receiving the PEP, and whether they discussed any of the training topics with other officers post-PEP. These circumstances will be considered as variables in our outcome analyses. Although the investigators expect change to occur in a linear manner (e.g., as more officers are trained fewer NSIs occur), the intervention effect could be curvilinear due to diffusion of information from trained to untrained officers. As such, the investigators will test for both linear and non-linear effects of time on the outcome.

Level 3: Although the investigators aim to shift police attitudinal norms about PWID, sex workers and HIV-positive persons and reduce adverse behaviors through a theory-driven framework (Aim 2), it is unrealistic to expect police to admit misconduct (e.g., physical or sexual abuse, soliciting bribes) to interviewers. Fortunately, the investigators are in the unique position of having, Proyecto El Cuete, a parallel cohort of PWID in Tijuana (Robertson, Garfein et al. 2014). Since 2010, 866 PWIDs have undergone semi-annual HIV tests and surveys including questions on police encounters. This includes negative experiences such as syringe confiscation, arrests near SEPs and drug treatment sites, sexual and physical abuse by police, as well as positive experiences, such as police referrals to SEPs or OST. The availability of these data enables us to externally assess the impact of the PEP on PWID risk behaviors by comparing PWIDs' policing experiences before vs. after PEP. Since El Cuete is funded through 2020, the investigators will have data pre-PEP, during the 2 years of PEP scale-up, and 2 years post-PEP. The investigators hypothesize a significant interaction between the PEP phase and Time, with the sharpest declines being observed during the post-PEP phase. The investigators will also create models with interview time (baseline, 6-months, 12-months, through 72-months) as the sole main fixed effect and introduce a quadratic term, as the investigators may observe a curvilinear trend due to the PEP over time. These findings and results from Proyecto ESCUDO will be used to inform cost-effectiveness analyses, using measures collected from both police and PWID in sensitivity analyses.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Active-duty police officer
* Completion of 3-hour PEP course
* Completion of the pre- and post-PEP surveys
* Follow-up consent
* For level 2: report encountering syringes within the last 6 months comprise the follow-up sampling frame

Exclusion Criteria:

* Did not complete 3-hour PEP course
* Did not complete pre- and post-PEP surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-05-29 (Actual); Study Completion 2018-05-29 (Actual)

PRIMARY OUTCOMES:
Incidence of Occupational Needle Stick Injuries | 3 years
  • The number of incident NSIs reported by each police officer, under the surveillance system. Cumulative NSI incidence will be measured over a three year period to accommodate the implementation of the step-wedge design intervention framework.

SECONDARY OUTCOMES:
HIV Knowledge | 0, 3, 6, 12, 18 and 24 months
  Knowledge score: knowledge of transmission, prevention and treatment of HIV and related infections (STIs and viral hepatitis).
Attitudinal and behavior changes | 0, 3, 6, 12, 18 and 24 months
  Attitudes score: attitudes towards PWID, sex workers and HIV-infected persons.
Adverse behaviors that interfere with HIV prevention | 0, 3, 6, 12, 18 and 24 months
  Self-reporting of adverse behaviors that interfere with HIV prevention (i.e. syringe confiscation and syringe-related arrests) and Tijuana police department geo-coded arrest data will be used to determine the rate of arrests that occur near SEP and drug treatment programs, pre- and post-PEP.
Protective behaviors | 2 years
  Self-reporting of protective behaviors for HIV prevention (i.e. use of gloves as barrier protection during pat-downs and arrests, self-reported reductions in syringe confiscation) and Tijuana police department geo-coded arrest data will be used to determine the extent to which the PEP decreases the number of arrests near SEP and OST sites in Tijuana, pre- and post-PEP.

OTHER OUTCOMES:
Mediating and moderating factors | 2 years
  Potential mediating and moderating factors influencing PEP efficacy from SDT constructs (motivation, years spent in the police force and autonomous support from supervisors) within each model used to assess the effect of the intervention of the outcome (e.g., NSI incidence).

CONTACTS AND LOCATIONS:
Overall Officials: Steffanie A Strathdee, PhD, Principal Investigator — Associate Dean of Global Health Sciences, Harold Simon Professor, Chief, Division of Global Public Health, University of California San Diego, Department of Medicine; Leo Beletsky, JD, MPH, Principal Investigator — Associate Professor of Law and Health Sciences, School of Law & Bouvé College of Health Sciences, Northeastern University, Adjunct Professor, Division of Global Public Health, University of California San Diego Department of Medicine
Locations (1):
- Instituto de Capacitacion Y Adiestramiento Profesional, Tijuana, Estado de Baja California, Mexico

REFERENCES:
- [Background] Strathdee SA, Arredondo J, Rocha T, Abramovitz D, Rolon ML, Patino Mandujano E, Rangel MG, Olivarria HO, Gaines T, Patterson TL, Beletsky L. A police education programme to integrate occupational safety and HIV prevention: protocol for a modified stepped-wedge study design with parallel prospective cohorts to assess behavioural outcomes. BMJ Open. 2015 Aug 10;5(8):e008958. doi: 10.1136/bmjopen-2015-008958. PMID 26260350
- [Derived] Baker P, Arredondo J, Borquez A, Clairgue E, Mittal ML, Morales M, Rocha-Jimenez T, Garfein R, Oren E, Pitpitan E, Strathdee SA, Beletsky L, Cepeda JA. Municipal police support for harm reduction services in officer-led referrals of people who inject drugs in Tijuana, Mexico. Harm Reduct J. 2021 Jul 26;18(1):76. doi: 10.1186/s12954-021-00513-4. PMID 34311765